CLINICAL TRIAL: NCT04182542
Title: Effects of Capacitive Radiofrequency at the Dermis and Adipose Tissue in the Abdominal Region
Brief Title: Effects of Capacitive Radiofrequency at the Dermis and Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Collaborators: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor/Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AN-010
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Adiposity; Abdominal Obesity
Keywords: Capacitive Radiofrequency; Abdominal Adipose Tissue
MeSH Terms: conditions — Obesity; Obesity, Abdominal | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know, when analyzing the samples, to which group they belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF (Experimental): The right side will be treated with radiofrequency
  Interventions: Device: Radiofrequency
- NI (No Intervention): The left side will not receive treatment.

INTERVENTIONS:
Device: Radiofrequency — The volunteers will receive radiofrequency (TECAR-BTL® device, with epidermal temperature above 40ºC) in the right infraumbilical abdominal region, with an application time of 10 minutes (2 minutes per applicator area) and the left region will be used as control. A single session will be held. After approximately 30 days of this application the material for histological analysis will be collected during the surgical act, at which point the skin and the subcutaneous tissue of the infraumbilical region are discarded by the surgeon.
  Other Names: Radiofrequency treatment
  Arms: RF

SUMMARY:
Noninvasive fat reduction is a rapidly expanding field of cosmetic rejuvenation, as many patients are unwilling to suffer the downtime and healing associated with traditional invasive liposuction. The radiofrequency (RF) device has been shown to be safe and effective for non-invasive fat reduction, as well as cutaneous enhancement and improvement of skin flaccidity (BOISNIC, et al., 2014).

DETAILED DESCRIPTION:
In Brazil, the search for satisfaction with self-image has been increasing, since the profile of the population has been altered by cultural factors such as industrialized foods with high caloric content and sedentary lifestyle. These factors result in the accumulation of adipose tissue in typical and atypical places, caused by the imbalance of the energy balance, that is, a higher caloric intake when compared to the energy consumption.

Noninvasive fat reduction is a rapidly expanding field of cosmetic rejuvenation, as many patients are unwilling to suffer the downtime and healing associated with traditional invasive liposuction. The radiofrequency (RF) device has been shown to be safe and effective for non-invasive fat reduction, as well as cutaneous enhancement and improvement of skin flaccidity (BOISNIC, et al., 2014).

Radiofrequency emits focused electromagnetic waves that find resistance in the tissue, generating heat (KRUEGUER, LEVY and SADICK, 2012). This thermal energy affects the triple helix structure of the collagen, subsequently breaking the intramolecular hydrogen bonds, resulting in immediate contraction of the collagen and neocollagenesis in the dermis, without interfering in the epidermis.

This neocollagenesis and remodeling of collagen results in a visibly compacted and organized dermis. Skin enhancement is an important effect, since patients that search for non-invasive fat reduction usually also seek improvement in skin flaccidity. This represents a substantial improvement over currently available technology (BOISNIC, et al, 2014).

There is controversy regarding the mechanism of fat mobilization. Some authors, after observing human skin cultures at the end of the series of RF treatments found a profound effect on subcutaneous adipocytes. The analysis resulted in altered morphology and increased expression of the pyroptosis marker, APAF-1, suggesting that pyroptosis induced by irreversible electroporation is the mechanism of action. Adipocyte pyroptosis results in the release of triglycerides from disintegrated cell membranes, but in a delayed and gradual manner, allowing a slow and safe removal through the interstitial space and liquid transport systems, lymphatic vessels and other metabolic functions. There was no evidence of necrosis or inflammatory changes observed in adipocytes after treatments with BodyFX, a type of radiofrequency (BOISNIC, et al, 2014).

Other authors say that the increase in temperature caused by RF has physiological effects, such as increased cellular metabolism, increased vasodilation and blood supply and activation of branches of the autonomic nervous system releasing adrenaline and noradrenaline (BELENKY, et al., 2012; PUMPRALA, et al., 2015, MESSINA, et al., 2017, RYDDEN and ARNER, 2017). These effects culminate in the better efficacy of lipolysis, which is a biochemical process where lipid hydrolysis occurs.

The evaluation and application of the protocol will be performed in the therapeutic resources laboratory of the physiotherapy course of Federal University of Triângulo Mineiro- UFTM (whose coordinator is the researcher responsible for this study), the material will be collected at the Clinical Hospital of the UFTM surgical center and the preparation and analysis of the slides will be carried out in the pathology laboratory of UFTM.

The women who will undergo plastic abdominoplasty surgery at the Clinical Hospital of the UFTM will be invited to participate in the study. These women are in the electronic queue awaiting surgery and will be invited by the plastic surgery team.

The volunteers will receive radiofrequency (TECAR-BTL® device, with epidermal temperature above 40ºC) in the right infraumbilical abdominal region, with an application time of 10 minutes (2 minutes per applicator area) and the left region will be used as control. A single session will be held. After approximately 30 days of this application the material for histological analysis will be collected during the surgical act, at which point the skin and the subcutaneous tissue of the infraumbilical region are discarded by the surgeon.

Fragments collected during surgery will be fixed in Methacarn (60% methanol, 30% chloroform, 10% acetic acid) for 2 hours at room temperature (RT). The slides will be made by the department of general pathology of the Federal University of the Triângulo Mineiro. Samples will be dehydrated in ethanol, diaphonized in xylol and embedded in paraffin. Histological sections of 5 μm thickness will be obtained in microtome (Jung) and placed on pre-coated sheets with polylysine. The histological sections will be stained with hematoxylin and eosin, Picro-sirius and Verhoeff. By the staining of Hematoxylin-Eosin will be analyzed the general morphology of the tissue including the quantity and volume of the adipose vacuoles, Picro-sirius the presence and morphology of the collagen fibers and Verhoeff the elastic fibers.

Blades stained by Hematoxylin-Eosin, Picro-sirius and Verhoeff will be visualized with a 20x objective. The images will be captured by a common light microscope and analyzed by the Axion Vision Automatic Image Analyzer System.

In this way the field to be quantified will be captured, photographed through a camera attached to the microscope and to the computer for image scanning. Images will be saved in TIFF format. All blade fields will be photographed and saved.

After the fields are saved, the Image J® program will be used to improve them, using the illumination reference so that they all have the same quality.

The percentage of collagen, elastic fibers and the analysis of the amount and volume of the adipose vacuole will be marked by the Image J® program and registered in a Microsoft Excel worksheet.

ELIGIBILITY:
Inclusion Criteria:

* Women who will undergo plastic abdominoplasty surgery at the Clinical Hospital of the Federal UFTM.

Exclusion Criteria:

* Sensitive and cognitive deficits
* Aged less than 18 years
* Metal implant at the application site
* Pacemakers
* Signs of infection
* Circulatory disorders
* Neoplasia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female submited to abdominal surgery
Enrollment: 20 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
percentage of collagen, elastic fibers and the analysis of the amount and volume of the adipose vacuole | 30 days
  The percentage of collagen, elastic fibers and the analysis of the amount and volume of the adipose vacuole will be marked by the Image J® program and registered in a Microsoft Excel worksheet- For the variables percentage of collagen, elastic fibers, number of fibroblasts and number of adipocytes will be performed the normality test with Shapiro Wilk. The paired t test will be used when data are normal and Wilcoxon when not normal. The differences observed will be considered significant when the probability of rejection of the null hypothesis is less than 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Adriana mendonça, Minas Gerais, Uberaba, Brazil

REFERENCES:
- [Background] Belenky I, Margulis A, Elman M, Bar-Yosef U, Paun SD. Exploring channeling optimized radiofrequency energy: a review of radiofrequency history and applications in esthetic fields. Adv Ther. 2012 Mar;29(3):249-66. doi: 10.1007/s12325-012-0004-1. Epub 2012 Feb 29. PMID 22382873
- [Background] Boisnic S, Divaris M, Nelson AA, Gharavi NM, Lask GP. A clinical and biological evaluation of a novel, noninvasive radiofrequency device for the long-term reduction of adipose tissue. Lasers Surg Med. 2014 Feb;46(2):94-103. doi: 10.1002/lsm.22223. PMID 24535760
- [Background] Krueger N, Levy H, Sadick NS. Safety and efficacy of a new device combining radiofrequency and low-frequency pulsed electromagnetic fields for the treatment of facial rhytides. J Drugs Dermatol. 2012 Nov;11(11):1306-9. PMID 23135079